CLINICAL TRIAL: NCT06015425
Title: Real-world Data Collection and Real-world Evidence Clinical Demonstration Study of tDCS for the Treatment of Depression in Perinatal Women
Brief Title: tDCS in Depression in Perinatal Women
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Seoul National University Hospital (Other)
Collaborators: Severance Hospital (Other); Ilsan Cha hospital (Other); Bundang CHA Hospital (Other); Ybrain Inc. (Industry)
Responsible Party: Principal Investigator, CHO HEE YOUNG, Professor, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HI23C0297
Record Dates: First submitted 2023-08-23; First posted 2023-08-29 (Actual); Last update posted 2023-08-31 (Actual); Status verified 2023-08

CONDITIONS: Depression; Pregnancy
Keywords: Transcranial Direct Current Stimulation; Depression; Pregnancy
MeSH Terms: conditions — Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- YMS-201B+ (Experimental): transcranial Direct Current Stimulation (tDCS) application 5 ~7 days a week for 4 weeks (total of 20~28 applications)
  Interventions: Device: MINDD STIM+

INTERVENTIONS:
Device: MINDD STIM+ — transcranial Direct Current Stimulation (tDCS) 2mA for 30 min; 30 sec of ramp-up and -down; left (anode) and right (cathode) Dorsolateral prefrontal cortex (DLPFC)

SUMMARY:
The goal of this clinical trial is Real-world data(RWD) collection and Real-world evidence(RWE) clinical demonstration study of Transcranial direct current stimulation(tDCS) for the treatment of depression in perinatal women. Participants will apply tDCS by themselves for 4 weeks at home. Researchers will compare Visit 1 to Visit 3 in one group.

DETAILED DESCRIPTION:
The prevalence of postpartum depression is known to be 10-20%, but the number of people who actually experience postpartum depression is reported to be higher. According to the 2018 survey on postpartum care by the Ministry of Health and Welfare(Korea), 50.3% of mothers experienced postpartum depression during the postpartum care period, and 33.9% of mothers aged 9 to 20 months postpartum were at risk of postpartum depression.

To this end, since the 1980s, safer and more effective depression methods such as tDCS and repetitive transcranial magnetic stimulation (rTMS), which are noninvasive brain stimulation methods using electricity and magnetism, have been developed. Research has begun as a treatment technique, and rTMS has been approved for depression by the US FDA in 2008 and the Ministry of Food and Drug Safety in Korea in 2013. It is becoming.

According to the report by Sreeraj (2016), tDCS monotherapy resulted in significant improvement in depressive and anxiety symptoms during pregnancy, and reported that it is likely to build an evidence base to strengthen the clinical usefulness of tDCS during pregnancy.

Therefore, through the actual use application of tDCS for the treatment of depression in perinatal women who are in the blind spot of drug treatment, RWD and RWE are collected.

ELIGIBILITY:
Inclusion Criteria:

* Patients with mild to moderate MDD among perinatal women aged between 19 and 50 years of age
* MDD refers to cases that clinically satisfy the diagnostic criteria for unipolar and nonpsychotic major depressive disorder according to the 5th edition of the Diagnostic and Statistical Manual of Mental Disorders (DSM-5).
* Mild and moderate symptoms are defined as non-severe conditions corresponding to a Beck Depression Inventory-II (BDI-II) score of 18 to 28 points or a Montgomery-Asberg Depression Rating Scale (MADRS) score of 14 to 34 points, which are the main evaluation variables.
* Those who can read and understand the subject explanation and consent form, and have Korean language proficiency at a level capable of responding to questionnaires
* In this study, since tDCS is not an absolute contraindication even for pregnant women, it is possible to participate in clinical demonstration studies unless the subject exclusion criteria are met.

Exclusion Criteria:

* Male
* Those who have been diagnosed with Post-Traumatic Stress Disorder (PTSD) or Obsessive Compulsive Disorder (OCD) among psychiatric comorbid anxiety disorders
* Those diagnosed with bipolar or psychotic major depressive disorder
* Among those diagnosed with Seizure Disorders, those who are judged by the clinician to be inappropriate for this clinical trial
* A person who scores 5 or more in MADRS question 10 (suicidal ideation)
* A person who has attempted suicide within 6 months from the date of screening or a person who, as determined by the clinician, has a suicide risk that requires hospitalization in a protective ward
* Those who are judged to have problems with EEG and DC stimulation electrode attachment due to scalp deformities, inflammatory reactions, or other dermatological problems
* A person who is judged to have other reasons for prohibiting the use of tDCS medical devices (refer to the example below)

  * A person who inserts a head metal plate
  * Users of implantable medical devices such as pacemakers and implantable cardioverter defibrillators.
  * Wearers of life-sustaining medical devices such as artificial heart lungs or users of implantable medical devices such as electrocardiographs
* Those who show clinically serious disorders in the cardiovascular system, digestive system, respiratory system, endocrine system, and central nervous system that affect the application and effectiveness evaluation of medical devices during the study period (e.g., those who have difficulty breathing while sitting still) If you have an endocrine system/central nervous system disease that is not controlled by medication, etc.)
* Those who participated in other clinical trials within 30 days from the date of screening
* Those who have applied transcranial direct current stimulation within 6 months from the date of screening
* In addition to the above, those who have clinically significant findings that are considered inappropriate for this clinical demonstration study as determined medically by the investigator or person in charge

Ages: 19 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Women who have a uterus and ovaries and are likely to become pregnant and give birth
Enrollment: 125 (Estimated)
Dates: Start 2023-10-01 (Estimated); Primary Completion 2024-03-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Korean-Beck Depression Inventory-II (K-BDI-II) score change for depressive symptoms | At 4 weeks after treatment
  Average change of K-BDI-II at 4 weeks after treatment compare to the base respectively. This scale contains 21 questions, each answer being scored on a scale value of 0 to 3. Higher total scores indicate more severe depressive symptoms.The lower the total score, the better the symptoms.
Montgomery-Åsberg Depression Rating Scale (MADRS) score change for depressive symptoms | At 4 weeks after treatment
  It is evaluated on 10 items, including outward sadness, spontaneously reported sadness, internal tension, sleep deprivation, loss of appetite, difficulty concentrating, laziness (boredom), loss of feeling, pessimistic thoughts, and suicidal thoughts. It is evaluated as ~6 points, and the total score is 0~60 points, and the change in score after 4 weeks is the Primary Outcome Measure.

SECONDARY OUTCOMES:
Center for Epidemiologic Studies Depression Scale (CESD-R) score change for depressive symptoms | At 4 weeks after treatment
  The CESD developed by Radloff et al. in 1977 for the evaluation of depressive symptoms was revised to reflect the diagnostic criteria for major depressive episodes in the DSM-IV (Eaton, 2004). Dysphoria, anhedonia, psychomotor retardation/agitation, suicide Items reflecting accidents have been added. Self-report 20-item scale, each item measured from 0 to 4 points and the change in score after 4 weeks is the Secondary Outcome Measures.
Korean Version of Edinburgh Postnatal Depression Scale (K-EPDS) score change for depressive symptoms | At 4 weeks after treatment
  It evaluates the symptoms experienced while experiencing postpartum depression rather than a general depression test. It was developed by Cox et al. in 1987 and adapted and standardized in Korea by Kim Yong-gu et al. in 2005. With a total score of 30, a score of 10 or more, the cut-off point, is evaluated as having depressive symptoms and the change in score after 4 weeks is the Secondary Outcome Measures.

OTHER OUTCOMES:
Actigraphy/Lifelog Service Use | At 4 weeks after treatment
  Tracking parameters such as sleep stages, score, mode, etc. And Evaluation using an application through CESD-R , previously developed by the research team.
Korean version of the Insomnia Severity Index (ISI-K) score change for Insomnia | At 4 weeks after treatment
  It is a questionnaire to evaluate the severity of insomnia and consists of a total of 7 questions. The total score ranges from 0 to 28, and a score of 15 or more, the cutoff point, is considered to be insomnia.
Korean version of Depression Anxiety Stress Scales-21 items (K-DASS-21) score change for Depression, anxiety, and stress | At 4 weeks after treatment
  It consists of a total of 21 questions, each with 7 questions for depression, anxiety, and stress, and the response to each question was selected from 0 points (not applicable at all) to 3 points (very much applicable). Each depression, anxiety, and stress subscore is obtained by summing up the scores of the corresponding items, and each score represents an individual's level of depression, anxiety, and stress.
Obstetric questionnaire. | At 4 weeks after treatment
  Obstetrics-related information was evaluated using questionnaires on general characteristics of pregnant women, pregnancy preparation questionnaires, and quarterly morning sickness questionnaires.

CONTACTS AND LOCATIONS:
Overall Officials: Hee Young Cho, Study Director — Seoul National University Hospital; san lee, Principal Investigator — Severance Hospital; Min-Kyoung Kim, Principal Investigator — Ilsan Cha hospital; Chun Il Park, Principal Investigator — Bundang CHA Hospital
Locations (1):
- Seoul National University Hospital, Seoul, Republic of Korea, South Korea

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Baran J, Leszczak J, Baran R, Biesiadecka A, Weres A, Czenczek-Lewandowska E, Kalandyk-Osinko K. Prenatal and Postnatal Anxiety and Depression in Mothers during the COVID-19 Pandemic. J Clin Med. 2021 Jul 20;10(14):3193. doi: 10.3390/jcm10143193. PMID 34300358
- [Background] Caparros-Gonzalez RA, Alderdice F. The COVID-19 pandemic and perinatal mental health. J Reprod Infant Psychol. 2020 Jul;38(3):223-225. doi: 10.1080/02646838.2020.1786910. No abstract available. PMID 32615801
- [Background] de Tychey C, Spitz E, Briancon S, Lighezzolo J, Girvan F, Rosati A, Thockler A, Vincent S. Pre- and postnatal depression and coping: a comparative approach. J Affect Disord. 2005 Apr;85(3):323-6. doi: 10.1016/j.jad.2004.11.004. PMID 15780702
- [Background] Grimm S, Beck J, Schuepbach D, Hell D, Boesiger P, Bermpohl F, Niehaus L, Boeker H, Northoff G. Imbalance between left and right dorsolateral prefrontal cortex in major depression is linked to negative emotional judgment: an fMRI study in severe major depressive disorder. Biol Psychiatry. 2008 Feb 15;63(4):369-76. doi: 10.1016/j.biopsych.2007.05.033. Epub 2007 Sep 21. PMID 17888408
- [Background] Hollins K. Consequences of antenatal mental health problems for child health and development. Curr Opin Obstet Gynecol. 2007 Dec;19(6):568-72. doi: 10.1097/GCO.0b013e3282f1bf28. PMID 18007135
- [Background] Kurzeck AK, Kirsch B, Weidinger E, Padberg F, Palm U. Transcranial Direct Current Stimulation (tDCS) for Depression during Pregnancy: Scientific Evidence and What Is Being Said in the Media-A Systematic Review. Brain Sci. 2018 Aug 14;8(8):155. doi: 10.3390/brainsci8080155. PMID 30110930
- [Background] Stein A, Gath DH, Bucher J, Bond A, Day A, Cooper PJ. The relationship between post-natal depression and mother-child interaction. Br J Psychiatry. 1991 Jan;158:46-52. doi: 10.1192/bjp.158.1.46. PMID 2015451
- [Background] Vigod S, Dennis CL, Daskalakis Z, Murphy K, Ray J, Oberlander T, Somerton S, Hussain-Shamsy N, Blumberger D. Transcranial direct current stimulation (tDCS) for treatment of major depression during pregnancy: study protocol for a pilot randomized controlled trial. Trials. 2014 Sep 18;15:366. doi: 10.1186/1745-6215-15-366. PMID 25234606
- [Background] Vigod SN, Murphy KE, Dennis CL, Oberlander TF, Ray JG, Daskalakis ZJ, Blumberger DM. Transcranial direct current stimulation (tDCS) for depression in pregnancy: A pilot randomized controlled trial. Brain Stimul. 2019 Nov-Dec;12(6):1475-1483. doi: 10.1016/j.brs.2019.06.019. Epub 2019 Jun 19. PMID 31257092
- [Background] Wu Y, Espinosa KM, Barnett SD, Kapse A, Quistorff JL, Lopez C, Andescavage N, Pradhan S, Lu YC, Kapse K, Henderson D, Vezina G, Wessel D, du Plessis AJ, Limperopoulos C. Association of Elevated Maternal Psychological Distress, Altered Fetal Brain, and Offspring Cognitive and Social-Emotional Outcomes at 18 Months. JAMA Netw Open. 2022 Apr 1;5(4):e229244. doi: 10.1001/jamanetworkopen.2022.9244. PMID 35486403
- [Background] Oh J, Jeon S, Ha TH, Myung W, Lee SH, Ko YH, Kim DH, Lee HY, Chae JH. Effect of Home-based Self-administered Transcranial Direct Stimulation in Patients with Mild to Moderate Major Depressive Disorder: A Single-arm, Multicentral Trial. Clin Psychopharmacol Neurosci. 2023 May 30;21(2):271-278. doi: 10.9758/cpn.2023.21.2.271. PMID 37119219
- [Background] Bikson M, Ganho-Avila A, Datta A, Gillick B, Joensson MG, Kim S, Kim J, Kirton A, Lee K, Marjenin T, Onarheim B, Rehn EM, Sack AT, Unal G. Limited output transcranial electrical stimulation 2023 (LOTES-2023): Updates on engineering principles, regulatory statutes, and industry standards for wellness, over-the-counter, or prescription devices with low risk. Brain Stimul. 2023 May-Jun;16(3):840-853. doi: 10.1016/j.brs.2023.05.008. Epub 2023 May 16. PMID 37201865
- [Background] Lorenzetti V, Allen NB, Fornito A, Yucel M. Structural brain abnormalities in major depressive disorder: a selective review of recent MRI studies. J Affect Disord. 2009 Sep;117(1-2):1-17. doi: 10.1016/j.jad.2008.11.021. Epub 2009 Feb 23. PMID 19237202
- [Background] Das S, Holland P, Frens MA, Donchin O. Impact of Transcranial Direct Current Stimulation (tDCS) on Neuronal Functions. Front Neurosci. 2016 Nov 30;10:550. doi: 10.3389/fnins.2016.00550. eCollection 2016. PMID 27965533
- [Background] Fregni F, Boggio PS, Nitsche MA, Marcolin MA, Rigonatti SP, Pascual-Leone A. Treatment of major depression with transcranial direct current stimulation. Bipolar Disord. 2006 Apr;8(2):203-4. doi: 10.1111/j.1399-5618.2006.00291.x. No abstract available. PMID 16542193
- [Background] Rigonatti SP, Boggio PS, Myczkowski ML, Otta E, Fiquer JT, Ribeiro RB, Nitsche MA, Pascual-Leone A, Fregni F. Transcranial direct stimulation and fluoxetine for the treatment of depression. Eur Psychiatry. 2008 Jan;23(1):74-6. doi: 10.1016/j.eurpsy.2007.09.006. Epub 2007 Nov 19. No abstract available. PMID 18023968
- [Background] Brunoni AR, Valiengo L, Baccaro A, Zanao TA, de Oliveira JF, Goulart A, Boggio PS, Lotufo PA, Bensenor IM, Fregni F. The sertraline vs. electrical current therapy for treating depression clinical study: results from a factorial, randomized, controlled trial. JAMA Psychiatry. 2013 Apr;70(4):383-91. doi: 10.1001/2013.jamapsychiatry.32. PMID 23389323